CLINICAL TRIAL: NCT00002250
Title: A Phase I Study of Recombinant Human CD4 Immunoglobulin G (rCD4-lgG) in Patients With HIV-Associated Immune Thrombocytopenic Purpura
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 076A; D0177g
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1991-08

CONDITIONS: Immune Thrombocytopenic Purpura ( ITP ); HIV Infections
Keywords: Recombinant Proteins; IgG; Drug Evaluation; Antigens, CD4
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; HIV Infections | interventions — CD4 Immunoadhesins

INTERVENTIONS:
Drug: CD4-IgG

SUMMARY:
To test the effectiveness of recombinant human CD4 Immunoglobulin G (CD4-IgG) in the treatment of HIV-associated immune thrombocytopenic purpura in patients with all levels of HIV infection.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Dapsone at a constant dose level and only as a prophylaxis for Pneumocystis carinii pneumonia (PCP).
* Zidovudine (AZT) at a constant dose for the 12 weeks of treatment, except if AZT-related toxicity is observed.

Patients must have the following:

* HIV seropositive (asymptomatic, AIDS-related complex, or AIDS).
* HIV-associated immune thrombocytopenic purpura.
* The ability to sign a written informed consent form, which must be obtained prior to treatment.
* A willingness to abstain from all other experimental therapy for HIV infection during the entire study period.
* Patients currently on zidovudine are not excluded. However, the zidovudine dose level must remain constant for 4 weeks prior to entry and for the 12 weeks of treatment, except if zidovudine related toxicity is observed.
* A life expectancy of at least 3 months.

Prior Medication:

Allowed:

* Dapsone at a constant dose for more than 2 weeks prior to study entry.
* Zidovudine at a constant dose for 4 weeks prior to study entry.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions and symptoms are excluded:

* Active serious opportunistic infection (excluding positive block cultures of Mycobacterium avium complex or Cytomegalovirus).
* Malignancies other than Kaposi's sarcoma.
* Tumor-associated edema.
* Visceral Kaposi's sarcoma.
* Significant neurologic, cardiac, or liver disease.

Concurrent Medication:

Excluded:

* Ganciclovir (DHPG). Pyrimethamine. Clindamycin. Sulfadiazine. Folinic acid. Prednisone. Intravenous gamma globulin. Intravenous acyclovir. Interferon. Systemic corticosteroids. Non-steroidal anti-inflammatory drugs (NSAIDs). Known immunomodulatory agents. Dideoxycytosine. Dideoxyinosine. Nucleoside analogs (with the exception of zidovudine or topical acyclovir). Any experimental therapy.

Patients with the following are excluded:

* Active serious opportunistic infection (excluding positive block cultures of Mycobacterium avium complex or Cytomegalovirus).
* Malignancies other than Kaposi's sarcoma.
* Kaposi's sarcoma requiring therapy.
* Tumor-associated edema.
* Visceral Kaposi's sarcoma.
* Significant neurologic, cardiac, or liver disease.
* Conditions requiring excluded concomitant medications.
* Herpes virus infection requiring intravenous acyclovir.

Prior Medication:

Excluded for a minimum of 4 weeks prior to study entry:

* Chemotherapy.
* Immunomodulatory agents.
* Any experimental therapy.

Prior Treatment:

Excluded for a minimum of 4 weeks prior to study entry:

* Radiation therapy.
* Any experimental therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- San Francisco Gen Hosp, San Francisco, California, United States

REFERENCES:
- [Background] Kahn J, Hassner A, Arri C, Coleman R, Kaplan L, Volberding P, Ammann A, Abrams D. A phase 1 study of recombinant human CD4 immunoglobulin g (rCD4-IgG) in patients with HIV-associated immune thrombocytopenic purpura. Int Conf AIDS. 1991 Jun 16-21;7(2):221 (abstract no WB2156)